CLINICAL TRIAL: NCT05980286
Title: Impact of Music Improvisation Training on Cognitive Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1R61AG073669 (NIH); 1R61AG073669 (NIH)
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Aging; Cognitive Aging; Cognitive Impairment; Cognitive Training; Cognitively Normal Older Adults; Mild Cognitive Impairment
Keywords: Aging; Brain Aging; Cognition; Cognitive Engagement; Mild Cognitive Impairment; Music; Music-based Intervention; Music Training; Older Adults
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: We will conduct a 2-arm randomized pilot trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piano Improvisation Training (Experimental): This intervention will involve group piano improvisation training sessions once a week for 12 weeks, in addition to daily in-home practice for 4-5 days.
  Interventions: Behavioral: Piano Improvisation
- Music Listening Training (Active Comparator): The music listening condition will involve group music listening sessions (led by a trained instructor) once a week for 12 weeks and daily in-home music listening practice.
  Interventions: Behavioral: Music Listening

INTERVENTIONS:
Behavioral: Piano Improvisation — Piano Improvisation taught by a professional instructor for 12 weeks.
  Arms: Piano Improvisation Training
Behavioral: Music Listening — Music Listening facilitated by a professional instructor for 12 weeks.
  Arms: Music Listening Training

SUMMARY:
This project will develop and test the effects and mechanisms of a music improvisation training intervention on self-regulation of older adults with and without MCI. The investigator's overall hypothesis is that improvisation training will lead to improvements in self-regulation, compared to controls, and that improvisation training will be associated with specific changes in prefrontal brain networks and ultimately cognitive engagement.

DETAILED DESCRIPTION:
Approximately 5.8 million adults age 60 and over in the United States live with Alzheimer disease and related dementias (AD/ADRD) at a cost of $290 billion per year. Older adults with mild cognitive impairment (MCI), an intermediate stage between typical aging and dementia, are 3-5 times more likely to progress to AD than those with normal cognition. Late-life engagement in cognitively challenging activities is associated with decreased risk of cognitive decline, and there is a need to address cognitive inactivity. Music interventions are a promising strategy to address late-life cognitive inactivity. Music training can change brain structure and function in non-musician adults, thereby leading to cognitive, perceptual, and psychosocial advantages. These changes in cognitive function are thought to occur because the multimodal, complex nature of music facilitates training-induced neural plasticity. However, the mechanisms are not yet understood, and most studies used traditional or rote keyboard training techniques. Music training based on improvisation principles-the spontaneous generation of musical melodies and rhythms-will likely have more potent effects on cognition and brain function. Improvisation facilitates cognitive flexibility, self-monitoring, novel idea generation, execution of unplanned motor sequences and entrance into a state of flow. Biologically, improvisation is associated with distinct neural patterns involving activation of prefrontal networks and other brain networks that are affected by aging. As a mechanism of behavior change, it is likely that improvisation training will uniquely improve self-regulation (the ability to monitor and control one's own behavior, emotions, or thoughts and modify to situational demands). Yet, no research has tested whether improvisation training can improve self-regulation and facilitate maintenance of cognitively challenging activities among older adults with and without MCI. This project will develop and test the effects and mechanisms of a music improvisation training intervention on self-regulation of older adults with and without MCI. Our overall hypothesis is that improvisation training will lead to improvements in self-regulation, compared to controls, and that improvisation training will be associated with specific changes in prefrontal brain networks and ultimately cognitive engagement. Our project has two phases. In the R61 phase, the study will develop a music improvisation training intervention that aims to improve self-regulation among older adults with and without MCI and conduct a 2-arm randomized pilot study to (i) examine feasibility and acceptability of the intervention and study methods and (ii) determine its effects on the hypothesized mechanism of self-regulation. If milestones are met, the study will proceed to the R33 phase and conduct a randomized mechanistic trial to examine the effects of the intervention, compared to an attention control, on self-regulation and cognitive engagement among older adults with and without MCI. The findings from this study will improve our understanding of the underlying mechanisms of how music training interventions can facilitate behavior change to maintain health of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and over
* Living independently in the community
* Sufficient visual and hearing acuity (age-related to normal hearing loss, with assistive devices) as measured by audiometer
* Less than three years of formal music training (as indicated by private music lessons does not include group or ensemble classes) and not currently reading or engaging in music performance
* English fluency rated fairly well to well
* Montreal Cognitive Assessment (MoCA) score of 22-30 or diagnosis of "mild cognitive impairment
* Not currently taking psychoactive medications, antidepressants, or sleep medications that could adversely affect cognitive abilities.

Exclusion criteria:

* Medical diagnosis of dementia (any etiology)
* Inability to move the hands or use all 10 digits (extensive arthritis, neuropathy, missing digits)
* Score < 22 on Montreal Cognitive Assessment (MoCA)
* Current (but not prior) severe psychiatric disorder, serious medical condition (e.g., stroke, TIA) that would interfere with participation in the study
* Poor English fluency
* Musician or previously trained in jazz improvisation, more than three years of formal music instruction or training and/or currently engaged in musical performance
* Plans to move out of the area within six months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julene Johnson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Department of Disability and Aging Services (DAS) Sites, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Piano Improvisation: This intervention will involve group piano improvisation training sessions once a week for 12 weeks, in addition to daily in-home practice for 4-5 days.
- Music Listening: The music listening condition will involve group music listening sessions (led by a trained instructor) once a week for 12 weeks and daily in-home music listening practice.
Period: Overall Study
Arm/Group | Piano Improvisation | Music Listening
Started | 24 | 29
Completed | 22 | 19
Not Completed | 2 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Piano Improvisation | Music Listening | Total
Number analyzed (Participants) | 24 | 29 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (5.8) | 75.9 (8.8) | 74.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 13 | 22
  White | 11 | 11 | 22
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 22 | 27 | 49
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants] — San Francisco County
  Participants
    United States | 24 | 29 | 53
Education [Count of Participants; unit: Participants] — Education: High school or less
  Participants | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Retention in Study
Description: This outcome is the proportion of participants who completed post-test assessments and remained in the study.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Piano Improvisation Training | Music Listening Training
Number analyzed (Participants) | 24 | 29
Participants | 22 | 21

2. Primary Outcome: Adherence to Intervention
Description: This outcome will document participant adherence to the intervention. The percentage of participants who completed at least 6 out of 12 sessions.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Piano Improvisation Training: This intervention will involve group piano improvisation training sessions once a week for 12 weeks, in addition to daily in-home practice for 4-5 days.Piano Improvisation: Piano Improvisation taught by a professional instructor for 12 weeks.
- Music Listening Training: The music listening condition will involve group music listening sessions (led by a trained instructor) once a week for 12 weeks and daily in-home music listening practice. Music Listening: Music Listening facilitated by a professional instructor for 12 weeks.
Arm/Group | Piano Improvisation Training | Music Listening Training
Number analyzed (Participants) | 24 | 29
Participants | 21 | 16

3. Primary Outcome: Satisfaction With Intervention
Description: This survey item was part of a longer feasibility and acceptability survey that was created for this study. This question measures the degree to which participants reported being satisfied with the intervention. This item was "Overall, how would you rate the quality of the sessions?" on a 5-point scale (1-poor, 2-fair, 3-good, 4-very good, or 5-excellent). Scores range from 1-5, with higher scores indicating better satisfaction. We report the percentage of participants who rated the intervention as good to excellent (scores of 3-5).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Piano Improvisation | Music Listening
Number analyzed (Participants) | 24 | 29
Participants | 24 | 27

4. Secondary Outcome: Short Self-Regulation Questionnaire
Description: The Short Self-Regulation Questionnaire is a 31-item measure of the ability to regulate behavior in order to achieve desired future outcomes. This is the short form of the Self-Regulation Questionnaire (SRQ) developed by Brown et al. in 1999. Each item was scored on a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The questionnaire scores range from 31 to 155, with higher scores indicating better self-regulation behavior.
Time Frame: Baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Piano Improvisation: This intervention will involve group piano improvisation training sessions once a week for 12 weeks, in addition to daily in-home practice for 4-5 days per week.
Arm/Group | Piano Improvisation | Music Listening
Number analyzed (Participants) | 24 | 29
units on a scale | -0.32 (10.02) | 0.95 (11.93)

5. Secondary Outcome: Florida Cognitive Activities Scale
Description: The Florida Cognitive Activities Scale is a self-report 25-item questionnaire (0-never to 5-daily) used to assess frequency of engagement in cognitive activity for older adults. A Total Cognitive Activity (TCA) score is calculated by summing scores on all 25 items, with scores ranging from 0-100. Higher scores indicate more frequent engagement in cognitive activity.
Time Frame: Baseline and 12-week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Piano Improvisation | Music Listening
Number analyzed (Participants) | 24 | 29
units on a scale | 0.86 (9.90) | -1.95 (12.04)

6. Secondary Outcome: National Institutes of Health ToolBox Self-Efficacy
Description: The NIH Toolbox Self-Efficacy Scale is a 10-item self-reported measure that assesses belief in one's capacity to manage and have control over meaningful events in life. Scores for each item range from 1 to 5 (never to very often) with scores ranging from 10-50. Higher scores indicate higher self-efficacy.
Time Frame: Baseline and 12-week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Piano Improvisation | Music Listening
Number analyzed (Participants) | 24 | 29
units on a scale | -0.50 (4.41) | -0.63 (5.06)

7. Secondary Outcome: Short Grit Scale
Description: The Short Grit Scale (Grit-S) is a self-report, 8-item questionnaire that measures the extent to which individuals are able to maintain focus and interest and persevere in obtaining long-term goals. The Short Grit Scale (Grit-S) retains the 2-factor structure of the original Grit Scale (Duckworth, Peterson, Matthews, & Kelly, 2007) with 4 fewer items and improved psychometric properties. Scores for each item range from 1 to 5, with overall scores being calculated by added up all points and dividing by 8. Scores range from 1-5. Higher scores indicate a higher level of "grit," or perseverance.
Time Frame: Baseline and 12-week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Piano Improvisation | Music Listening
Number analyzed (Participants) | 24 | 29
units on a scale | -0.86 (3.62) | -0.74 (2.40)

8. Secondary Outcome: Five Facets of Mindfulness
Description: Measures components of mindfulness, which is a tendency to attend to the present moment with a non-judgemental attitude. Scores for each item range from 1 to 5 (never to always true), with higher scores representing lower non-judgemental attitude.The Total FFMQ can be divided by 39 to get an average item score. Total score ranges from 39 to 195, and higher scores suggest a better mindful self-awareness.
Time Frame: Baseline and 12-week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Piano Improvisation | Music Listening
Number analyzed (Participants) | 24 | 29
units on a scale | 0.23 (5.36) | 0.79 (4.73)

ADVERSE EVENTS:
Time Frame: up to 14 weeks, which represented the week when the baseline assessment was done, the 12-week intervention, and the week when the post-intervention assessment was done.
Description: Adverse events were graded from mild to severe.Potential mild adverse effects while completing a questionnaire could include boredom, fatigue, frustration, and loss of confidentiality. Potential mild adverse events related to piano improvisation training may include frustration, stress, and mild musculoskeletal fatigue. Moderate adverse events may include the falls and moderate musculoskeletal fatigue or pain. Severe adverse events might include cardiovascular events and death.
Arm/Group | Piano Improvisation | Music Listening
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/29
Other Adverse Events (participants affected / at risk) | 4/24 | 2/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Piano Improvisation (N=24) | Music Listening (N=29)
Musculoskeletal fatige (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Two participants experienced pain in the hands during keyboard practice
Frustration with learning new skill (General disorders) | 2 (2) | 0 (0) — Two participants experienced frustration with learning a new skill
Frustration with participants' attendance (General disorders) | 0 (0) | 2 (2) — Two participants expressed frustration with participants who missed intervention sessions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT05980286/Prot_SAP_000.pdf